CLINICAL TRIAL: NCT00143494
Title: The Estimation of Abdominal Pressure by the Bladder and Gastric Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Davide Chiumello, Policlinico Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1200
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Critically Ill Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Critically hill, mechanically ventilated patients
  Interventions: Procedure: measurement of abdominal pressure

INTERVENTIONS:
Procedure: measurement of abdominal pressure — measurement of abdominal pressure with different volume and saline temperature

SUMMARY:
The investigators aim to compare the bladder pressure to the gastric pressure in critically ill patients.

DETAILED DESCRIPTION:
In critically ill patients, we will measure the gastric pressure by a gastric balloon and the bladder pressure by the intra-vesical pressure to find the optimal method to estimate the abdominal pressure.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients during invasive mechanical ventilation

Exclusion Criteria:

* Contraindication to measure the bladder pressure

Ages: 16 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-07; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To estimate the bladder pressure | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: davide chiumello, MD, Principal Investigator — Policlinico Hospital
Locations (1):
- Policlinico Hospital, Milan, Italy

REFERENCES:
- [Result] Chiumello D, Tallarini F, Chierichetti M, Polli F, Li Bassi G, Motta G, Azzari S, Carsenzola C, Gattinoni L. The effect of different volumes and temperatures of saline on the bladder pressure measurement in critically ill patients. Crit Care. 2007;11(4):R82. doi: 10.1186/cc6080. PMID 17655744